CLINICAL TRIAL: NCT01275807
Title: Acupuncture as an Integrated Intervention for the Control of Symptoms of Climacteric Syndrome in Patients Affected by Breast Cancer
Brief Title: Effectiveness and Safety of Acupuncture for Climacteric Syndrome in Patients With Breast Cancer
Acronym: AcCliMaT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Usl di Bologna (Other Government)
Collaborators: Regione Emilia-Romagna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DGR-2025/2008-Lesi
Record Dates: First submitted 2010-12-30; First posted 2011-01-12 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Climacteric Syndrome
Keywords: climacteric, climacteric syndrome
MeSH Terms: interventions — Acupuncture Therapy; Medicine, Chinese Traditional; Self Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- acupuncture (Experimental): 10 acupuncture sessions
  Interventions: Device: acupuncture
- self care (Active Comparator): psychological support, phisical exercice, diet, self care groups
  Interventions: Other: self care

INTERVENTIONS:
Device: acupuncture — 10 sessions of acupuncture
  Other Names: chinese traditional medicine
  Arms: acupuncture
Other: self care — physical exercice, diet, self help groups, psychological support
  Other Names: self help
  Arms: self care

SUMMARY:
The purpose of the investigators study is to create the evidence of effectivness on climacteric syndrome in patients affected by breast cancer, by acupuncture added to the standard care (self care).

DETAILED DESCRIPTION:
The study will be performed under randomized, open, controlled design. The effect of acupuncture and control group will be compared including the following outcomes: Greene climacteric scale score, quality of life (MenQol italian version), overall improvement in climacteric syndrome, adverse effects from treatment.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer
* thermoregulation symptoms from at least 6-8 weeks - at least 6 hot flushes a day
* climateric simptoms
* age from 18 to 65 years
* spontaneous or caused by chemotherapy amenorrea
* hormone therapy for breast cancer
* Green climateric scale score = or > of 15
* performance status Eastern Cooperative Oncology Group (ECOG) < or = to 1
* the patient agrees to follow physical exercice
* diet and self-help groups

Exclusion Criteria:

* Hormone substitutive Therapy (TOS) during the last month
* other systemic treatments for climateric syndrome (tibolone, antidepressants, homeopathy)
* chemotherapy or radiotherapy
* patients who refuses acupuncture

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2010-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Greene climacteric scale | baseline ( 14 days before randomization) , between the 5th and 6th session af acupunture(only for experimental arm) at 14 weeks after randomization and at 3 and at 6 month after randomization for both arms.
  Greene's score as measure for severity of menopausal symptoms. Change in the number of hot flashes.

CONTACTS AND LOCATIONS:
Overall Officials: grazia lesi, MD, Study Director — Bologna Local Health District - Azienda Usl di Bologna
Locations (4):
- Italy (4):
  - Unità operativa (U.O.) salute donna infanzia e adolescenza e Unità operativa Consultori, Bologna, Bologna
  - Oncologic Medicine, Carpi Hospital, Carpi, Modena
  - Dipartimento Anestesia, rianimazione, terapia del dolore e comparto operatorio,, Piacenza
  - U.O. Medicina Oncologica - Ospedale Santa Maria Nuova Reggio Emilia, Reggio Emilia

REFERENCES:
- [Background] Gupta P, Sturdee DW, Palin SL, Majumder K, Fear R, Marshall T, Paterson I. Menopausal symptoms in women treated for breast cancer: the prevalence and severity of symptoms and their perceived effects on quality of life. Climacteric. 2006 Feb;9(1):49-58. doi: 10.1080/13697130500487224. PMID 16428125
- [Derived] Lesi G, Razzini G, Musti MA, Stivanello E, Petrucci C, Benedetti B, Rondini E, Ligabue MB, Scaltriti L, Botti A, Artioli F, Mancuso P, Cardini F, Pandolfi P. Acupuncture As an Integrative Approach for the Treatment of Hot Flashes in Women With Breast Cancer: A Prospective Multicenter Randomized Controlled Trial (AcCliMaT). J Clin Oncol. 2016 May 20;34(15):1795-802. doi: 10.1200/JCO.2015.63.2893. Epub 2016 Mar 28. PMID 27022113